CLINICAL TRIAL: NCT00105651
Title: A Smoking, Alcohol, and Depression Intervention for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IIR 98-500
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Combined nursing invention

INTERVENTIONS:
Behavioral: Combined nursing invention

SUMMARY:
Data from the Surveillance, Epidemiology and End Results (SEER) cancer registry indicates that head and neck cancers (HN Ca) are nearly twice as common in veterans as non-veterans. HN Ca patients are at an increased risk for smoking, alcohol consumption and depression, all of which contribute to a further decline in their quality of life (QoL). In the HN Ca population, diagnosis and treatment of smoking, alcohol intake and depression are sub-optimal, thereby affecting QoL and survival. Numerous studies have documented that smoking, alcohol and depression are interrelated and research on multi-modal interventions has been suggested.

DETAILED DESCRIPTION:
Background:

Data from the Surveillance, Epidemiology and End Results (SEER) cancer registry indicates that head and neck cancers (HN Ca) are nearly twice as common in veterans as non-veterans. HN Ca patients are at an increased risk for smoking, alcohol consumption and depression, all of which contribute to a further decline in their quality of life (QoL). In the HN Ca population, diagnosis and treatment of smoking, alcohol intake and depression are sub-optimal, thereby affecting QoL and survival. Numerous studies have documented that smoking, alcohol and depression are interrelated and research on multi-modal interventions has been suggested.

Objectives:

To determine whether a combined intervention for smoking, alcohol intake, and depression improves the QoL of veterans with HN Ca.

Methods:

Patients from three VA medical centers (Ann Arbor, MI; Dallas, TX; Gainesville, FL) who have at least one of the three disorders of smoking, drinking and depression were randomized to either usual care or the combined intervention. Data was collected on smoking, alcohol consumption, depression and QoL at baseline, 6- and 12- months after the intervention (or non-intervention). The main analyses consisted of analysis of covariance (ANCOVA) to compare the scores on the SF-36 mental health scores and on the emotional domain of Head and Neck Quality of Life Questionnaire between the experimental and control group at 6- and 12- month follow up. Additional analyses examineded smoking, alcohol intake, and depression scores at these same time points.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Head and Neck Cancer patients who: 1) screen positive for at least one of the three health problems of smoking, alcohol and depression; 2) are not pregnant; 3) are greater than 18 years of age; and 4) speak english. Exclusion criteria include patients who: 1) have metastatic disease (terminal); or 2) have unstable psychiatric/mental conditions such as suicidal ideation, acute psychosis, severe alcohol dependence or dementia.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A. Duffy, PhD MS RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Larry Myers, MD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

REFERENCES:
- [Result] Lambert MT, Terrell JE, Copeland LA, Ronis DL, Duffy SA. Cigarettes, alcohol, and depression: characterizing head and neck cancer survivors in two systems of care. Nicotine Tob Res. 2005 Apr;7(2):233-41. doi: 10.1080/14622200500055418. PMID 16036280
- [Result] Taylor JC, Terrell JE, Ronis DL, Fowler KE, Bishop C, Lambert MT, Myers LL, Duffy SA, Bradford CR, Chepeha DB, Hogikyan ND, Prince ME, Teknos TN, Wolf GT; University of Michigan Head and Neck Cancer Team. Disability in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 2004 Jun;130(6):764-9. doi: 10.1001/archotol.130.6.764. PMID 15210560
- [Result] Cheng SS, Terrell JE, Bradford CR, Ronis DL, Fowler KE, Prince ME, Teknos TN, Wolf GT, Duffy SA. Variables associated with feeding tube placement in head and neck cancer. Arch Otolaryngol Head Neck Surg. 2006 Jun;132(6):655-61. doi: 10.1001/archotol.132.6.655. PMID 16785412
- [Result] Terrell JE, Ronis DL, Fowler KE, Bradford CR, Chepeha DB, Prince ME, Teknos TN, Wolf GT, Duffy SA. Clinical predictors of quality of life in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 2004 Apr;130(4):401-8. doi: 10.1001/archotol.130.4.401. PMID 15096421
- [Result] Duffy SA, Terrell JE, Valenstein M, Ronis DL, Copeland LA, Connors M. Effect of smoking, alcohol, and depression on the quality of life of head and neck cancer patients. Gen Hosp Psychiatry. 2002 May-Jun;24(3):140-7. doi: 10.1016/s0163-8343(02)00180-9. PMID 12062138
- [Result] Duffy SA, Jackson FC, Schim SM, Ronis DL, Fowler KE. Racial/ethnic preferences, sex preferences, and perceived discrimination related to end-of-life care. J Am Geriatr Soc. 2006 Jan;54(1):150-7. doi: 10.1111/j.1532-5415.2005.00526.x. PMID 16420213
- [Result] Duffy SA, Ronis DL, Valenstein M, Fowler KE, Lambert MT, Bishop C, Terrell JE. Depressive symptoms, smoking, drinking, and quality of life among head and neck cancer patients. Psychosomatics. 2007 Mar-Apr;48(2):142-8. doi: 10.1176/appi.psy.48.2.142. PMID 17329608
- [Result] Duffy SA, Ronis DL, Valenstein M, Lambert MT, Fowler KE, Gregory L, Bishop C, Myers LL, Blow FC, Terrell JE. A tailored smoking, alcohol, and depression intervention for head and neck cancer patients. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2203-8. doi: 10.1158/1055-9965.EPI-05-0880. PMID 17119047
- [Result] Duffy SA, Ronis D, Fowler K, Schim SM, Jackson FC. Differences in veterans' and nonveterans' end-of-life preferences: a pilot study. J Palliat Med. 2006 Oct;9(5):1099-105. doi: 10.1089/jpm.2006.9.1099. PMID 17040147
- [Result] Karvonen-Gutierrez CA, Ronis DL, Fowler KE, Terrell JE, Gruber SB, Duffy SA. Quality of life scores predict survival among patients with head and neck cancer. J Clin Oncol. 2008 Jun 1;26(16):2754-60. doi: 10.1200/JCO.2007.12.9510. PMID 18509185